CLINICAL TRIAL: NCT00065247
Title: Beat Osteoporosis: Nourish and Exercise Skeletons (BONES)
Brief Title: The BONES Project: Building Healthy Bones in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: R01HD037752 (NIH)
Record Dates: First submitted 2003-07-18; First posted 2003-07-22 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-06

CONDITIONS: Osteoporosis
Keywords: Bone; Children; After-school program; Osteoporosis; Calcium; Physical activity
MeSH Terms: conditions — Osteoporosis; Motor Activity

INTERVENTIONS:
Behavioral: Beat Osteoporosis: Nourish and Exercise Skeletons (BONES) Project

SUMMARY:
The Beat Osteoporosis: Nourish and Exercise Skeletons (BONES) Project is an after-school program that includes weight loading physical activity, nutrition and bone health education, and calcium-rich snacks. The program is designed to improve bone health in early elementary school children.

DETAILED DESCRIPTION:
Osteoporosis is a serious public health concern expected to threaten 52 million Americans by the year 2010. This debilitating disease comes at an annual cost of $17 billion. By optimizing bone development during the growing years, individuals can lower their risk of osteoporosis by building an adequate reserve of bone. This study will implement and evaluate an after-school program with exercise, education, and diet components designed to improve bone quality and muscle strength in early elementary school children.

First and second grade children from 84 after school programs in 33 diverse communities throughout Massachusetts and Rhode Island will be enrolled in the study. After-school programs will be randomized to either the BONES Project, to the BONES Project plus a parent/caregiver component, or to a no-intervention control group. The BONES curriculum will be implemented 4 days per week over a 20- to 25-week period; each after-school program will implement the program for 2 years. Participants will be followed for an additional year, assuming they remain in the after-school program or do not withdraw for some other reason. All parents will be asked to complete a Child Medical History survey and a Parent Health Survey at baseline, during the 2-year intervention, and at the end of the follow-up year. Parents in the BONES Project plus parent/caregiver component will receive a newsletter and worksheet 5 times per year.

Participants will be assessed by quantitative ultrasound, height, weight, and body composition measurements, muscular strength, self competence, physical activity level, food knowledge and preference, calcium intake, perceived parental support, and sleep habits.

ELIGIBILITY:
Inclusion Criteria

* Enrolled in participating after-school program
* Live in Massachusetts or Rhode Island

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1500
Dates: Start 1999-06; Study Completion 2004-05

CONTACTS AND LOCATIONS:
Overall Officials: Christina D. Economos, PhD, Principal Investigator — Tufts University
Locations (1):
- Tufts University Gerald J. and Dorothy R. Friedman School of Nutrition, Science and Policy, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Economos CD, Hennessy E, Chui K, Dwyer J, Marcotte L, Must A, Naumova EN, Goldberg J. Beat osteoporosis - nourish and exercise skeletons (BONES): a group randomized controlled trial in children. BMC Pediatr. 2020 Feb 21;20(1):83. doi: 10.1186/s12887-020-1964-y. PMID 32093625